CLINICAL TRIAL: NCT00797498
Title: A Clinical Outcomes Protocol of Photon/Proton Beam Radiation Therapy for Cancers of the Nasal Cavity and/or Paranasal Sinuses
Brief Title: Photon/Proton Radiation Therapy for Cancers of the Nasal Cavity and/or Paranasal Sinuses
Acronym: SI01
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0604-SI01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Cancers of Nasal Cavity; Cancers of Paranasal Sinuses
Keywords: Nasal Cavity; Paranasal Sinuses; Proton Radiation; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xerostomia Questionnaire: All of the tests, procedures and treatments may be considered standard of care for someone with this type of cancer, except for the Xerostomia Questionnaire.
  Interventions: Other: Xerostomia questionnaire

INTERVENTIONS:
Other: Xerostomia questionnaire — All of the tests, procedures and treatments may be considered standard of care for someone with this type of cancer, except for the Xerostomia Questionnaire.

SUMMARY:
The purpose of this study is to collect information from a questionnaire and medical records to see what effects proton radiation has on cancer and collect and analyze morbidity outcomes: incidence of Xerostomia (dry mouth) and tumor control.

DETAILED DESCRIPTION:
The study is non interventional outcomes protocol designed to collect information from a questionnaire and medical records to see what effects proton radiation has on cancer and collect and analyze morbidity outcomes: incidence of Xerostomia (dry mouth) and tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of nasal cavity and/or paranasal sinuses.
* Will receive treatment with proton radiation.

Exclusion Criteria:

* Evidence of distant metastasis.
* Previous radiation for head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Radiation Oncology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2006-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Grade 3 or higher of xerostomia Incidence of Xerostomia | One year after the end of radiation therapy.

SECONDARY OUTCOMES:
Collect and analyze tumor control outcomes | When each patient has been followed for a minimum of 12 months with final analysis after 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD, MS, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Korzeniowski S, Reinfuss M, Skolyszewski J. The evaluation of radiotherapy after incomplete surgery in patients with carcinoma of the maxillary sinus. Int J Radiat Oncol Biol Phys. 1985 Mar;11(3):505-9. doi: 10.1016/0360-3016(85)90181-6. PMID 2982772
- [Background] Shidnia H, Hornback NB, Saghafi N, Sayoc E, Lingeman R, Hamaker R. The role of radiation therapy in the treatment of malignant tumors of the paranasal sinuses. Laryngoscope. 1984 Jan;94(1):102-6. doi: 10.1002/lary.5540940119. PMID 6690866
- [Background] Ellingwood KE, Million RR. Cancer of the nasal cavity and ethmoid/sphenoid sinuses. Cancer. 1979 Apr;43(4):1517-26. doi: 10.1002/1097-0142(197904)43:43.0.co;2-b. PMID 445347
- [Background] Gadeberg CC, Hjelm-Hansen M, Sogaard H, Elbrond O. Malignant tumours of the paranasal sinuses and nasal cavity. A series of 180 patients. Acta Radiol Oncol. 1984;23(2-3):181-7. doi: 10.3109/02841868409136009. PMID 6331089
- [Background] Lavertu P, Roberts JK, Kraus DH, Levine HL, Wood BG, Medendorp SV, Tucker HM. Squamous cell carcinoma of the paranasal sinuses: the Cleveland Clinic experience 1977-1986. Laryngoscope. 1989 Nov;99(11):1130-6. doi: 10.1288/00005537-198911000-00005. PMID 2811551
- [Background] Paulino AC, Marks JE, Bricker P, Melian E, Reddy SP, Emami B. Results of treatment of patients with maxillary sinus carcinoma. Cancer. 1998 Aug 1;83(3):457-65. PMID 9690538
- [Background] Myers LL, Nussenbaum B, Bradford CR, Teknos TN, Esclamado RM, Wolf GT. Paranasal sinus malignancies: an 18-year single institution experience. Laryngoscope. 2002 Nov;112(11):1964-9. doi: 10.1097/00005537-200211000-00010. PMID 12439163
- [Background] Waldron JN, O'Sullivan B, Gullane P, Witterick IJ, Liu FF, Payne D, Warde P, Cummings B. Carcinoma of the maxillary antrum: a retrospective analysis of 110 cases. Radiother Oncol. 2000 Nov;57(2):167-73. doi: 10.1016/s0167-8140(00)00256-5. PMID 11054520
- [Background] Jiang GL, Morrison WH, Garden AS, Geara F, Callender D, Goepfert H, Ang KK. Ethmoid sinus carcinomas: natural history and treatment results. Radiother Oncol. 1998 Oct;49(1):21-7. doi: 10.1016/s0167-8140(98)00075-9. PMID 9886693
- [Background] Parsons, J.T., Mendenhall, W.M., Stringer, S.P., Cassisi, N.J. & Million, R.R.: Nasal cavity and paranasal sinuses. In: Perez CA, Brady LW, eds. Principles and practice of radiation oncology, 3rd ed. Lippincott-Raven Publishers, Philadelphia; 1997, p. 941-959.
- [Background] Katz TS, Mendenhall WM, Morris CG, Amdur RJ, Hinerman RW, Villaret DB. Malignant tumors of the nasal cavity and paranasal sinuses. Head Neck. 2002 Sep;24(9):821-9. doi: 10.1002/hed.10143. PMID 12211046
- [Background] Le QT, Fu KK, Kaplan M, Terris DJ, Fee WE, Goffinet DR. Treatment of maxillary sinus carcinoma: a comparison of the 1997 and 1977 American Joint Committee on cancer staging systems. Cancer. 1999 Nov 1;86(9):1700-11. PMID 10547542
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation optic neuropathy after megavoltage external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):755-63. doi: 10.1016/0360-3016(94)90346-8. PMID 7960976
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation retinopathy after external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):765-73. doi: 10.1016/0360-3016(94)90347-6. PMID 7960977
- [Background] Bhandare N, Monroe AT, Morris CG, Bhatti MT, Mendenhall WM. Does altered fractionation influence the risk of radiation-induced optic neuropathy? Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1070-7. doi: 10.1016/j.ijrobp.2004.12.009. PMID 15990010